CLINICAL TRIAL: NCT07332403
Title: The Relationship Between Diaphragm Function Assessed by Ultrasound and Weaning Success in Mechanically Ventilated Patients in the ICU
Acronym: ICU
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berfin Seyrek, Resident Physician in Anesthesiology and Reanimation, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMICUWEAN
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Weaning Mechanical Ventilation; Ultrasonography; Intensive Care (ICU); Assesment of Diaphragmatic Function by Ultrasound to Predict Weaning Success in Mechanical Ventilated Intensive Care Unit Patients; Diaphragm Usg
Keywords: weaning; diaphragm usg; succesful weaning; unsuccesful weaning; diaphragm excursion; ıwı

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diaphragm ultrasound before weaning procedure — Using the ultrasound device, diaphragmatic usg was performed by an experienced clinician and the investigator. A linear probe was placed on the chest wall along the right anterior and mid-axillary lines at the 8-9th intercostal spaces over the zone of apposition and B-mode imaging was used to visualize the right hemidiaphragm as a three-layered structure: two parallel echogenic lines with a hypoechoic layer in between. Diaphragmatic thickness at end-inspiration(TEI) and end-expiration(TEE) was measured during the patient's spontaneous breathing. Three measurements were obtained, and the mean value was calculated. The diaphragmatic thickening fraction (DTF) was then calculated using the formula. Subsequently, a convex probe was placed at the right subcostal midclavicular line along the costal margin, and diaphragmatic motion was assessed using M-mode ultrasonography.Diaphragmatic excursion amplitude was measured, with three measurements obtained and the mean value recorded.

SUMMARY:
The diaphragm is the most important muscle involved in the respiratory system and is solely responsible for approximately 65-80% of vital capacity. When it contracts, it increases the volume of the thoracic cavity, leading to a decrease in intrathoracic pressure and allowing airflow from the atmosphere into the alveoli. Diaphragmatic atrophy begins as early as the first hours of mechanical ventilation (MV). Animal studies have demonstrated that prolonged mechanical ventilation results in diaphragmatic dysfunction, a condition defined as ventilator-induced diaphragmatic dysfunction (VIDD). Ultrasonographic evaluation of the diaphragm has shown a 32% reduction in diaphragmatic strength within the first 72 hours.

Assessment of diaphragmatic function is crucial for predicting weaning success. Ultrasonography (USG) is a practical, safe, non-invasive, bedside method that provides real-time results and allows both morphological and functional evaluation of the diaphragm. The ability to assess diaphragmatic contraction simultaneously enables measurement and follow-up of diaphragmatic thickness. This is also clinically useful for diagnosing diaphragmatic dysfunction and diaphragmatic paralysis.

The aim of this study was to evaluate the relationship between diaphragmatic function assessed by ultrasonography and weaning success in intubated patients followed in the intensive care unit.

In patients admitted to the Intensive Care Unit who received invasive mechanical ventilation for at least 24 hours, were included in the study, were considered ready for the weaning process by the attending clinician independently of the study protocol, and had adequate cognitive function, the following parameters were measured by the investigator prior to separation from mechanical ventilation while the patient was in spontaneous breathing mode (pressure support ventilation, PSV): respiratory rate, minute ventilation, tidal volume, maximal inspiratory pressure (MIP), rapid shallow breathing index (RSBI), airway occlusion pressure at 100 ms (P0.1), PaO₂/FiO₂ ratio, PaCO₂, integrated weaning index (IWI), and static and dynamic lung compliance.

After a 30-minute stabilization period, the planned procedures were explained to the patient, and the head of the bed was elevated to 30 degrees. Using the ultrasound device routinely employed in our clinic, diaphragmatic ultrasonography was performed by an experienced clinician and the investigator. A linear probe was placed on the chest wall along the right anterior and mid-axillary lines at the 8th-9th intercostal spaces over the zone of apposition, and B-mode imaging was used to visualize the right hemidiaphragm as a three-layered structure consisting of two parallel echogenic lines (the diaphragmatic pleura and the peritoneal membrane) with a hypoechoic structure in between (the muscle itself).

Diaphragmatic thickness at end-inspiration (TEI) and end-expiration (TEE) was measured during the patient's spontaneous breathing. Three measurements were obtained, and the mean value was calculated. Using these mean values, the diaphragmatic thickening fraction (DTF) was calculated according to the formula:

DTF = [(TEI - TEE) / TEE] × 100.

Subsequently, a convex probe was placed at the right subcostal midclavicular line along the costal margin, and diaphragmatic motion was visualized using M-mode ultrasonography. Diaphragmatic excursion amplitude was measured, with three measurements obtained and the mean value recorded.

Patients who successfully completed a 30-minute spontaneous breathing trial (SBT) in PSV mode were extubated. Weaning was considered successful in patients who were able to maintain spontaneous breathing for 48 hours without mechanical ventilatory support. Patients who maintained effective spontaneous breathing without mechanical support for more than 48 hours were classified as the successful weaning group, whereas those who required reintubation and a return to mechanical ventilation at any point during the weaning process were classified as the unsuccessful weaning group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were admitted to the Intensive Care Unit of Fatih Sultan Mehmet Training and Research Hospital between March 2025 and December 2025, received invasive mechanical ventilation for at least 24 hours, and were considered ready for separation from mechanical ventilation by the intensive care physician.
2. Patients aged 18 years and older.
3. Patients who provided written informed consent.

Exclusion Criteria:

1. Patients younger than 18 years of age.
2. Patients with a tracheostomy, neuromuscular disease, diaphragmatic paralysis, or spinal cord injury above the T8 level.
3. Patients with pneumothorax, pneumomediastinum, or chest wall and/or diaphragmatic injury.
4. Patients for whom informed consent could not be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the Intensive Care Unit of Fatih Sultan Mehmet Training and Research Hospital between March 2025 and December 2025, received invasive mechanical ventilation for at least 24 hours, and were considered ready for separation from mechanical ventilation by the intensive care physician.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
ultrasound assesment of Diaphragmatic function in patients undergoing weaning | Measurements were performed 30 minutes after patients were initiated on a spontaneous breathing trial following the decision to proceed with weaning.
  Measurement of diaphragmatic thickness and diaphragmatic excursion amplitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No